CLINICAL TRIAL: NCT02932397
Title: Efficacy of an Intravenous Dose of Propofol Versus Placebo in the Prevention of Coughing During Emergence of General Anesthesia Under Desflurane
Brief Title: Efficacy of Propofol vs Placebo in the Prevention of Coughing During Emergence of General Anesthesia Under Desflurane
Acronym: PROPOREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CE16.176
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Elective Surgery; Coughing
Keywords: Ambulatory surgery; Perioperative outcomes; General anesthesia under desflurane; Prevention of coughing; Propofol
MeSH Terms: conditions — Cough | interventions — Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): Active drug given to patients as an intravenous dose of 0.5 mg/kg of propofol
  Interventions: Drug: Intravenous dose of 0.5 mg/kg of propofol
- Saline solution (Placebo Comparator): Placebo drug given to patients as an intravenous dose of 0.05 mL/kg of saline solution (NaCl 0.9%)
  Interventions: Drug: Intravenous dose of 0.05 mL/kg of saline solution

INTERVENTIONS:
Drug: Intravenous dose of 0.5 mg/kg of propofol
  Arms: Propofol
Drug: Intravenous dose of 0.05 mL/kg of saline solution
  Arms: Saline solution

SUMMARY:
Emergence of general anesthesia is a critical period, in the same way as the induction of anesthesia, during which several adverse events may occur. Extubation may even be more difficult than the intubation, with a higher respiratory complications rate. Among these, cough is common and expected. It can be associated with significant complications including hypertension, tachycardia, increased intracranial pressure, bleeding at the surgical site or even wound dehiscence.

The incidence of coughing during emergence of general anesthesia varies depending on the type of airway instrumentation, the population under study, agents used for the maintenance of the anesthesia and techniques used to prevent coughing. In the literature, the incidence of coughing during emergence of general anesthesia under endotracheal intubation varies from 38 to 96%. In our center, the incidence of coughing during emergence of general anesthesia under desflurane and endotracheal intubation is 30 % according to a local preliminary study.

Propofol is well-known to inhibit airway reflexes. Total intravenous anesthesia (TIVA) is associated with a lower incidence of coughing compared to inhalated anesthesia. The efficacy of propofol at a subhypnotic dose to reduce coughing during emergence has recently been demonstrated in patients undergoing nasal surgery under sevoflurane. However, the most effective antitussive dose remains unknown and its efficacy during anesthesia under desflurane has not yet been demonstrated.

Propofol is rapidly available, simple to administer and has an interesting pharmacological profile, among others due to its short half-life.

The aim of this study is to evaluate if an intravenous bolus of 0.5 mg/kg of propofol is more effective than placebo administration to decrease the incidence of coughing during emergence of general anesthesia under desflurane (PROPOREV). Propofol could also reduce the incidence of postoperative nausea and vomiting (PONV).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 to 80 years undergoing elective surgery under general anesthesia with an orotracheal intubation;
* Patients of American Society of Anesthesiologists (ASA) I to III inclusively at the preoperative evaluation
* Patients affiliated to a medical insurance system.

Exclusion Criteria:

1. Ear, nose and throat (ENT) surgery, thoracic and neurological surgery ;
2. Participation refusal;
3. Patient allergic to or presenting a contraindication to propofol;
4. Patient with a tracheostomy;
5. Chronic coughing, i.e. daily cough for 8 weeks or more;
6. Asthma / severe or exacerbated chronic obstructive pulmonary disease (COPD);
7. Recent respiratory tracts infection (< 4 weeks);
8. Hemostasis disorders;
9. Patient known for a non-secure cerebral aneurysm;
10. Patient known for a difficult intubation (grade 3 or 4);
11. Patient suffering from mental, neurological, or severe cardiovascular disease;
12. Pregnant or breastfeeding women;
13. Patients with deafness and/or unable to have conversations in a normal voice;
14. Patient with language barrier (not speaking French, nor English);
15. Patient suffering from dementia or patient under guardianship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of coughing (between discontinuation of desflurane and minimum alveolar concentration (MAC) of 0.15 of desflurane) | one day, perioperative period
  Incidence of coughing during emergence of general anesthesia (between discontinuation of desflurane and MAC of 0.15 of desflurane) and its severity based on a 4-grade scale

SECONDARY OUTCOMES:
Incidence of coughing (between discontinuation of desflurane, MAC of 0.1 and 0.2 of desflurane, at extubation, as well as 5 and 10 min after extubation) | one day, perioperative period
  Incidence of coughing during emergence of general anesthesia (between MAC of 0.15 of desflurane and until 10 min after extubation) and its severity based on a 4-grade scale
Extubation time | one day, perioperative period
  Interval between discontinuation of desflurane and extubation
Sedation of the patient | one day, perioperative period
  Sedation of the patient two, five and ten minutes following extubation, then at 15 minutes interval in the recovery room, based on the Observer's Assessment of Alertness/Sedation Scale (OAA/A), until 30 minutes after the admission in the recovery room
Incidence of hypoventilation | one day, perioperative period
  incidence of hypoventilation (breathing rate < 8/min)
Incidence of hypoxic episode | one day, perioperative period
  incidence of hypoxic episode (oxygen saturation < 90%)
Blood pressure | one day, perioperative period
  Measurement of blood pressure before the induction and during emergence (every 5 min) in order to calculate incidence of fluctuation of non invasive blood pressure and heart rate of more than 20% between the values before induction of anesthesia until 10 min after extubation
Heart rate | one day, perioperative period
  Measurement of heart rate before the induction and during emergence (every 5 min) in order to calculate incidence of fluctuation of non invasive blood pressure and heart rate of more than 20% between the values before induction of anesthesia until 10 min after extubation
Agitation of the patient during emergence | one day, perioperative period
  Note the possible agitation of the patient during emergence
Complications | one day, perioperative period
  Describe potential complications secondary to the bolus of the substance under study at the emergence
Cumulative incidence of nausea/vomiting | one day, perioperative period
  Calculate cumulative incidence of nausea/vomiting between extubation and 30 minutes after the admission in the recovery room
Swallowing pain scores | one day, perioperative period
  Evaluate swallowing pain scores evaluated using a verbal simple numeric scale (0 = no pain et 10 = worst pain imaginable) 30 min after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Beaulieu, MD, PhD, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ouellet MF, Moore A, Williams S, Girard F, Desroches J, Ruel M, Beaulieu P. Efficacy of a propofol bolus against placebo to prevent cough at emergence from general anesthesia with desflurane: a randomized controlled trial. Can J Anaesth. 2023 May;70(5):842-850. doi: 10.1007/s12630-023-02401-w. Epub 2023 Feb 24. PMID 36829104